CLINICAL TRIAL: NCT03215771
Title: Longitudinal Observation of Myoelectric Upper Limb Orthosis Use Among Veterans With Upper Limb Impairment
Brief Title: Myoelectric Upper Limb Orthosis Use by Persons With TBI and Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Louis Stokes VA Medical Center (U.S. Federal Agency); Myomo (Industry)
Responsible Party: Principal Investigator, Stefania Fatone, PhD, BPO(Hons), Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-16-1-0733
Record Dates: First submitted 2017-07-03; First posted 2017-07-12 (Actual); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Traumatic Brain Injury; Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MyoPro + Motor Learning-Based Therapy (Experimental): Subjects received 9 weeks of motor learning-based therapy in combination with use of MyoPro myoelectric elbow wrist hand orthosis, followed by 9 weeks of home use with a customized exercise program.
  Interventions: Device: MyoPro Motion-G; Other: Motor Learning-Based Therapy

INTERVENTIONS:
Device: MyoPro Motion-G — The MyoPro Motion-G is an elbow-wrist-hand myoelectric orthosis.
Other: Motor Learning-Based Therapy — Motor learning-based (MLB) therapy included movement practice as close to normal as possible, high repetition, progression of challenge, part versus whole task practice, and knowledge of results. Treatment was customized to abilities of each subject and consisted of both MyoPro training and MLB therapy without device. Training with device was progressed using a hierarchy of challenge to increase complexity of movement. MLB therapy without device followed the same hierarchy, incorporating training of movements that could not be accomplished with the device and those that were trained with device. Movement quality was monitored and training practice was incrementally progressed as subject demonstrated improved ability to perform a given task/movement component. Subjects performed a custom home exercise program (HEP) on non-clinic days, increasing repetition as tolerated. At conclusion of in-clinic phase, individuals transitioned to a home phase where they continued to use the HEP.

SUMMARY:
The objective of this study was to document longitudinal outcomes in persons with traumatic brain injury (TBI) or stroke using the myoelectric upper limb orthosis with powered elbow and grasp in conjunction with motor learning-based therapy using both patient centric performance and patient reported outcome measures. Longitudinal observation allowed the investigators to detect both the initial therapeutic effects as well as the later functional outcomes of orthosis use. The investigators planned to recruit 15 Veterans and non-veterans who had TBI or stroke and upper limb impairment. The study required 29 visits over 22 weeks and was divided into three parts: orthotic fitting, therapy/training (9 weeks), and home use (9 weeks). Therapeutic and functional benefits were evaluated every 2 to 3 weeks over 18 weeks using simple, short clinical tests.

DETAILED DESCRIPTION:
This study had two aims: (1) to evaluate therapeutic and neuroplastic effects of a myoelectric upper limb orthosis in conjunction with motor learning-based therapy and (2) to evaluate the functional effects of a myoelectric upper limb orthosis in conjunction with motor learning-based therapy. The investigators planned to recruit 15 Veterans and non-veterans who had Traumatic Brain Injury (TBI) or stroke and upper limb impairment, were over 18 years of age and a minimum of 6 months from injury. The study required 29 visits over 22 weeks and was divided into three parts: orthotic fitting, therapy/training (9 weeks), and home use (9 weeks). Therapeutic and functional benefits were evaluated every 2 to 3 weeks over 18 weeks using simple, short clinical tests.

Subjects were enrolled in the study if they met eligibility criteria assessed at a screening visit. Once enrolled subjects were fit with a custom fabricated MyoPro Motion-G elbow-wrist-hand orthosis following standard clinical procedures. This process required up to three visits to cast, trial fit and deliver the orthosis. Subjects then participated in a standard-of-care motor learning based therapy protocol in conjunction with the PERL ("Push Eat Reach Lift") training program recommended by Myomo, which consists of a 9 week, 18 session training plan. Every second week, there was one session that combined therapy/training and outcomes evaluation.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* minimum 6 months since injury
* elbow, forearm, wrist and hand have full motion with little resistance from muscles when moved by someone else
* some ability to actively move the shoulder
* able to generate consistent and detectable electrical signals from the upper arm and forearm muscles
* able to read and comprehend the English language
* able to follow two-stage command
* cognitive abilities sufficient to perform testing and training protocols
* able to tolerate functional tasks for 60 minutes without excessive fatigue
* medically and psychologically stable
* at home support from a family member or care giver if needed

Exclusion Criteria:

* elbow, forearm, wrist and hand have less than full motion with high resistance from muscles when moved by someone else
* shoulder instability, pain or dislocation
* unable to safely support the weight of arm with added weight of the device without pain
* less than 12 weeks since botulinum toxin injection in the impaired arm
* new therapies/medications planned during study period
* skin rash or open wound on impaired arm
* inability to detect light touch or pain on impaired arm
* involuntary movements of the impaired arm
* pain or hypersensitivity in the impaired arm
* inability to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pundik S, McCabe J, Skelly M, Salameh A, Naft J, Chen Z, Tatsuoka C, Fatone S. Myoelectric Arm Orthosis in Motor Learning-Based Therapy for Chronic Deficits After Stroke and Traumatic Brain Injury. Front Neurol. 2022 Feb 8;13:791144. doi: 10.3389/fneur.2022.791144. eCollection 2022. PMID 35211080

RESULTS

PARTICIPANT FLOW:
Groups:
- MyoPro + Motor Based Learning: Subjects received 9 weeks of motor based therapy in combination with use of MyoPro myoelectric elbow wrist hand orthosis, followed by 9 weeks of home use with a customized exercise program.
  MyoPro Motion-G: The MyoPro Motion-G is an elbow-wrist-hand myoelectric orthosis.
Period: Overall Study
Arm/Group | MyoPro + Motor Based Learning
Started | 16
Stroke Subjects | 8
TBI Subjects | 8
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- MyoPro + Motor Based Learning: Subjects received 9 weeks of motor based therapy in combination with use of MyoPro myoelectric elbow wrist hand orthosis, followed by 9 weeks of home use with a customized exercise program.
  MyoPro Motion-G: The MyoPro Motion-G is a custom-fabricated elbow-wrist-hand myoelectric orthosis.
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.62 (19.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment of Motor Recovery for Upper Limb (FMA)
Description: Evaluation of motor impairment of the upper limb. Thirty-three items of movement coordination and reflex activity are scored with a 3-point Likert scale (0-66 points total) where higher scores represent less arm impairment.
Time Frame: Change in Fugl-Meyer Assessment of Motor Recovery for Upper Limb (FMA) from Baseline at Week 18
Population: combined results from 6 TBI and 7 stroke subjects
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- MyoPro + Motor Based Learning: Subjects received 9 weeks of motor based therapy in combination with use of MyoPro myoelectric elbow wrist hand orthosis, followed by 9 weeks of home use of the MyoPro along with a home exercise program.
  MyoPro Motion-G: The MyoPro Motion-G is an elbow-wrist-hand myoelectric orthosis.
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
score on a scale | 7.5 [5.4 to 9.7]

2. Secondary Outcome: Modified Ashworth Scale
Description: Using a 6-point scale, the clinician evaluates resistance to passive movement about a joint with varying degrees of velocity as follows:
  0 No increase in muscle tone.
  1 Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension.
  1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM.
  2 More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved.
  3 Considerable increase in muscle tone, passive movement difficult.
  4 Affected part(s) rigid in flexion or extension. A lower score represents less resistance to passive movement.
Time Frame: Change in Modified Ashworth Scale from Baseline at Week 18
Population: combined results from 6 TBI and 7 stroke subjects
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
score on a scale | -2.3 [-2.9 to -1.7]

3. Secondary Outcome: Chedoke Arm and Hand Activity Inventory (CAHAI)
Description: Used to assess performance of activities of daily living (ADLs). Measure consists of 13 functional tasks scores and the score for each functional task are summed to compute the total score. Scoring of each task is based on a 7-point scale (1=unable; 7=normal performance; minimum score is 13 points; maximum score is 91 points), where higher scores represent better performance of ADLs.
Time Frame: Change in Chedoke Arm and Hand Activity Inventory (CAHAI) from Baseline at Week 18
Population: combined results from 6 TBI and 7 stroke subjects
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
score on a scale | 8.8 [6.2 to 11.4]

4. Secondary Outcome: Orthotic and Prosthetic Users' Survey Satisfaction Module (OPUSsat)
Description: An 11-item patient-reported survey that assesses satisfaction with device using a 5-point Likert scale. Satisfaction with device is the sum of the scores (score range: 11-55), where higher scores indicate better satisfaction with device.
Time Frame: Change in Orthotic and Prosthetic Users' Survey satisfaction module (OPUSsat) from Baseline at Week 18
Population: combined results from 6 TBI and 7 stroke subjects
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
score on a scale | 26.7 [15.9 to 37.6]

5. Secondary Outcome: Craig Handicap Assessment and Rehabilitation Technique (CHART)
Description: A life-role participation survey measuring the level of handicap using objectively observable behaviors in five dimensions: physical, social, cognitive, mobility, and occupation. Survey responses are combined using formulas for each domain. The score in each domain is capped at 100 (total score range: 0-500). Higher scores represent better self-reported participation.
Time Frame: Change in Craig Handicap Assessment and Rehabilitation Technique (CHART) from Baseline at Week 18
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MyoPro + Motor Based Learning
Number analyzed (Participants) | 13
score on a scale | 34.9 [5.3 to 64.5]

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- MyoPro + Motor Based Learning: Subjects received 9 weeks of motor based therapy in combination with use of MyoPro myoelectric elbow wrist hand orthosis.
  MyoPro Motion-G: The MyoPro Motion-G is an elbow-wrist-hand myoelectric orthosis.
Arm/Group | MyoPro + Motor Based Learning
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03215771/Prot_SAP_000.pdf